# Clinical Investigation Plan (CIP)



Parent Procedure:



Additional Notes: Not applicable

Date 18 Oct 2023

# Approval:



### **Table of Contents**

| 1. | Clinical | Trial Summary Information | 7 |
|---|---|---|---|
| 2. | Identific | cation and Description of the Investigational Device | 12 |
| 3. | Justific | ation for the Design of the clinical investigation | 13 |
| | 3.1. | Synopsis | 13 |
| | 3.2. | Literature Review | 13 |
| | 3.3. | Pre-Clinical Testing | 15 |
| | 3.4. | Previous Clinical trial | 15 |
| | 3.5. | Justification for Administration | 17 |
| 4. | Benefits | s and Risks of the investigational device, clinical procedure and clinical investigation | 17 |
| | 4.1. | Anticipated benefits | 17 |
| | 4.2. | Risks associated with participation in the clinical investigation | 17 |
| | 4.3. | Possible interactions with concomitant medical treatments | 17 |
| | 4.4. | Steps that will be taken to control or mitigate risks | 17 |
| | 4.5. | Rationale for benefit-risk ratio | 17 |
| <b>5</b> . | Objectiv | ves & Hypotheses of the clinical investigation | 18 |
| | 5.1. | - · | |
| | 5. | 1.1. Patient participant objective | 18 |
| | 5. | 1.2. Partner participant objective | 18 |
| | 5.2. | Hypotheses | 18 |
| | | 2.1. Patient participant hypothesis | |
| | 5. | 2.2. Partner participant hypothesis | 18 |
| | 5.3 | Endpoints | 18 |
| | | 3.1.1. Patient Participant Endpoints | |
| | 5. | 3.1.2. Partner Participant Endpoints | 18 |
| | 5.4. | Methods and Timing for assessing, recording and analysing variables | 20 |
| | 5.5. | Equipment used for assessing clinical investigation variables and arrangements for monitori maintenance and calibration | ing |
| | 5.6. | Procedures for the replacement of participants | |
| | 5.7. | Investigation sites | |
| | | 7.1. Definition of completion of clinical investigation | |
| | 5.8. | Investigational device(s) and comparator(s) | 21 |
| 6. | Particip | ants | 22 |
| | 6. | 1.1. Inclusion criteria for participants selection | 22 |
| | 6. | 1.2. Exclusion criteria for participants selection | 22 |
| | 6. | 1.3. Criteria and procedures for patients withdrawal / lost to follow-up | 23 |
| | 6. | 1.4. Point of Enrolment | 23 |
| | 6. | 1.5. Total expected duration of the clinical investigation | 24 |

| | 6. | 1.6. Expected duration of each participant | 24 |
|---|---|---|---|
| | 6. | 1.7. Number of subjects & Distribution of enrolment across sites | 24 |
| | 6. | 1.8. Estimated time to reach enrolment number | 24 |
| | 6. | 1.9. Information on vulnerable, pregnant / breastfeeding population (if applicable) | 24 |
| 7. | | ıres | |
| | 7. | 1.1. Clinical-Investigation Procedures | 27 |
| | | Roles and Responsibilities | |
| | 7. | 2.1. Activities performed by sponsor representatives | 31 |
| | 7. | 2.2. Known / foreseeable factors affecting clinical investigation outcome or interpretation of results | 31 |
| | 7. | 2.3. Methods for addressing known / foreseeable factors | 32 |
| | 7. | 2.4. Follow-up period during clinical investigation | 32 |
| | | 2.5. Medical care for participants after completion of clinical investigation | |
| | 7. | | |
| | 7.3. | Monitoring Plan | 32 |
| 8. | Statistic | al Design and Analysis | 35 |
| | 8.1.<br>8. | Data Collection | |
| | 8.2. | Sample size calculation and justification | |
| | 8.3. | Pass / Fail Criteria | 36 |
| | 8.4. | Management of Controls and Bias | 37 |
| | 8.5. | Unused or spurious data (including drop-outs) management | 38 |
| 9. | Data Ma | nagement | 38 |
| | 9.1. | Methods (e.g. CRF) for data entry and collection | 38 |
| | 9.2. | Procedures used for handling CRF data | 38 |
| | 9.3. | Procedures for verification, validation and securing of electronic data systems (if applicable) | 38 |
| | 9.4. | Procedures to maintain and protect participant privacy | 38 |
| | 9.5. | Methods for database locking (start of analysis and storage) upon completion of clinical investigation | 38 |
| | 9.6. | Procedures for data retention | 38 |
| | 9.7. | Specified retention period | |
| | 9.8. | Other aspects of clinical quality assurance (As appropriate) | 39 |
| 10. | Amendr | nents to the CIP | 39 |
| 11. | Deviation | ns from clinical investigation plan (CIP) | 39 |
| | 11.1. | Exceptions that allow deviations to the CIP | 39 |
| | 11.2. | Procedures for recording, reporting and analysing CIP deviations | 39 |
| | 11.3. | Notification requirements and time-frames | 39 |
| 12. | Device A | Accountability | 40 |
| | 12.1. | Description of procedures for accountability of investigational devices | 40 |
| | 12.2. | Procedures for the return of investigational devices | 40 |



F&P , US, 2023



| 13. | Statements of Compliance | 40 |
|---|---|---|
| | 13.1. Conducting the investigation in accordance with the Declaration of Helsinki | 40 |
| | 13.2. Conducting this clinical investigation in compliance with regional or national regulations | 40 |
| | 13.3. Approval / Favourable opinion from the EC / Regulatory authority | 41 |
| | 13.4. Additional requirements imposed by the EC / Regulatory authority | 41 |
| | 13.5. Insurance for subjects | 41 |
| | 13.6. Financing of the clinical investigation | 41 |
| 14. | Informed Consent Process | 41 |
| | 14.1. General process for obtaining informed consent | 41 |
| | 14.2. Circumstances where informed consent cannot be gained | 41 |
| 15. | Adverse Events, Adverse device effects and device deficiencies | 42 |
| | 15.1. List of non-reportable events | 42 |
| | 15.2. Time period of reporting AEs & ADEs | 43 |
| | 15.3. Process for reporting AEs | 43 |
| | 15.4. Process of reporting DDs | 43 |
| | 15.5. Emergency contact details for reporting SAEs and SADEs | 43 |
| 16. | Suspension or premature termination of clinical investigation | 44 |
| | 16.1. Criteria and arrangements for suspension or premature termination | 44 |
| | 16.2. Criteria to assess and to break blinding/masking code | 44 |
| | 16.3. Requirements for follow-up and continued care | 44 |
| 17. | Publication Policy | 45 |
| | 17.1. Registration of clinical investigation in a publicly accessible database | 45 |
| | 17.2. Availability of clinical investigation results | 45 |
| 18. | Regulatory and Other References | 45 |
| | 18.1. Internal References | 45 |
| | 18.2. External References | 45 |
| | 18.3. Bibliography | 47 |
| 19. | Revision history | 48 |
| 20. | Appendix A – | |
| | 7.ppenaix.7. | |



F&P US, 2023

| Term | Abbreviation | Definition |
|---|---|---|
| Adverse event | AE | Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, including an abnormal laboratory finding, in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational device. |
| | | See also serious adverse event. |
| Apnea-Hypopnea<br>Index | АНІ | Measure of sleep apnea severity calculated from the number of apneic and hypopneic episodes combined per hour of sleep which last more than 10 seconds and are associated with a decrease in blood oxygenation <sup>1</sup> . |
| Auto-titrating<br>positive airway<br>pressure | APAP | Mode of non-invasive ventilation during which a low set pressure is supplied to the airway, unless an obstruction is detected, in which case pressure ramps up to a higher level, up to a set maximum limit. <sup>2,3</sup> |
| Bilevel positive airway pressure | BPAP | Mode of non-invasive ventilation during which two distinct pressure, one on inhalation and the other on exhalation, are supplied to the airway <sup>3</sup> . |
| | | A |
| Clinical<br>Investigation Plan | CIP | A document(s) that state the rationale, objectives, design and proposed analysis, methodology, monitoring, conduct and record-keeping of the clinical investigation. This is synonymous with Protocol. |
| Clinical Master<br>Data | CMD | Collates the body of knowledge related to the therapy and clinical procedures by documenting therapy background, and the latest clinical literature search strategy, results, and conclusions. |
| Case Report<br>Form/ electronic<br>Case Report Form | CRF/eCRF | Deidentified document used by the sponsor of a clinical investigation to record source information relating to a study subject, including investigational data which is collected, procedures that are followed, and adverse events that occur. This can be physical or stored on an electronic server. |
| Design History File | DHF | Compilation of documentation that describes the design history of a medical device. |
| Delegation of<br>Authority | DoA | This document will define, establish and allocate all investigation related duties and functions. |
| Design Review | DR | A milestone in the product development process whereby a design is evaluated against its requirements in order to verify outcomes of previous activities or identify issues. |
| Ethics Committee | EC | An independent body whose responsibility it is to review a Clinical Investigation in order to protect the rights, safety and wellbeing of participating human subjects. This is synonymous with Institutional Review Board (IRB). |
| Excessive<br>Daytime<br>Sleepiness | EDS | Subjective difficulty in maintaining an awake state, accompanied by increased ease of falling asleep when sedentary <sup>4</sup> . |



F&P

US, 2023

| Term | Abbreviation | Definition |
|---|---|---|
| Epworth<br>Sleepiness Scale | ESS | A widely used scale in the field of sleep medicine as a subjective measure of a patient's sleepiness. The scale estimates whether you are experiencing excessive sleepiness that possibly requires medical attention. |
| Fisher & Paykel<br>Healthcare | F&P | Fisher & Paykel Healthcare Ltd. |
| Good Clinical<br>Practice | GCP | A standard for the design, conduct, performance, monitoring, auditing, recording, analysis and reporting of Clinical Investigations that provides assurance that the data and reported results are credible and accurate, and that the rights, integrity and confidentiality of Investigation subjects are protected. Forms an integral part of ISO 14155:2020. |
| Investigators<br>Brochure | IB | A compilation of the clinical and non-clinical data on the investigational medical device(s) which is relevant to the Clinical Investigation. |
| Informed Consent<br>Form | ICF | A document that captures that the potential subject has discussed and understands what is being proposed by the clinical investigation and what is expected of them if they decide to sign the form and continue into the clinical investigation. Informed consent procedures are defined by the clinical investigation plan. |
| International<br>Council for<br>Harmonization | ICH | International body comprised of representatives from various national standards organizations, and intended to promote worldwide proprietary, industrial, and commercial standards. |
| Instructions For<br>Use | IFU | Also known as UI (user instructions); A document supplied with the investigational product that outlines how to use, clean, assemble and disassemble the investigational product. It also contains any relevant warnings and cautions and additional information about the operating requirements of the investigational product. |
| Institutional<br>Review Board | IRB | See also Ethics Committee (EC) |
| Good Clinical<br>Practice | GCP | A standard for the design, conduct, performance, monitoring, auditing, recording, analysis and reporting of Clinical Investigations that provides assurance that the data and reported results are credible and accurate, and that the rights, integrity and confidentiality of Investigation subjects are protected. Forms an integral part of ISO 14155:2020. |
| General Safety<br>and Performance<br>Requirements | GSPR | Set of requirements/product characteristics which are considered by the European authorities as being essential to ensuring that any new device will be safe and perform as intended throughout its life. |
| Non-invasive<br>Ventilation | NIV | Airway support administered through a mask wherein inhaled gases are supplied with positive end-expiratory pressure, often at a set tidal volume and rate. <sup>5</sup> |
| Obstructive Sleep<br>Apnea | OSA | Sleep-related breathing disorder characterized by recurrent interruptions in breathing during sleep due to temporary obstruction of the airway by lax, excessively bulky, or malformed pharyngeal tissues, with resultant hypoxemia and chronic lethargy <sup>6</sup> . |
| Obesity<br>Hypoventilation<br>Syndrome | OHS | Sleep-related disorder accompanied by severe overweightness, hypoxemia during sleep, and hypercapnia during the day, resulting from excessively slow or shallow breathing <sup>7</sup> . |



RP US, 2023

Doc. No:

Revision: A

| Term | Abbreviation | Definition |
|---|---|---|
| Positive Airway<br>Pressure | PAP | Mode of respiratory ventilation during which compressed air is supplied to the lungs to prevent episodes of airway collapse and to facilitate normal breathing <sup>3</sup> . |
| Principal/Primary<br>Investigator | PI | The qualified individual responsible for conducting the Clinical Investigation at an investigational site. |
| Protocol Deviation<br>Form | PDF | The record of all diversions from the procedures outlined in the clinical investigation plan. |
| Recruitment Script | RS | A standardized text delegated recruiters for the clinical investigation to use during the recruitment phase of the trial to ensure full disclosure of important points and consistency across staff. |
| Serious adverse event | SAE | Any adverse event that led to any of the following: Death Serious deterioration in the health of the subject, that resulted in any of the following: Life-threatening illness or injury Permanent impairment of a body structure or a body function Hospitalization or prolongation of patient hospitalization Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function Fetal distress, fetal death or a congenital physical or mental impairment or birth defect See also adverse event |
| Serious Adverse<br>Event Form | SAEF | A record of all serious adverse events and required additional analysis and review. Each serious adverse event is required to have its own completed serious adverse event form. |
| | N/A | |
| | N/A | |

# 1. Clinical Trial Summary Information

| Information | Details |
|---------------------------------|--------------|
| Clinical Investigation Details | |
| Title of Clinical Investigation | F&P US, 2023 |



&P US, 2023 Doc. No: Revision:

| Information | Details |
|---|---|
| Clinical Investigation<br>Description | This clinical investigation is designed to validate and confirm the overall performance and acceptability, of the F&P |
| Clinical Investigation<br>Device(s) used | PAP therapy, both in clinical settings and in-home environments for the treatment of various respiratory conditions, including obstructive sleep apnea (OSA). The F&P will be offered similarly to existing products on the market. |



F&P \_\_\_\_\_, US, 2023

| Information | Details |
|---|---|
| Inclusion / Exclusion | |
| Criteria(s) | Inclusion criteria: |
| | <ul> <li>Persons who are ≥22 years of age</li> </ul> |
| | <ul> <li>Persons who weigh ≥66 pounds (or 30 kg)</li> </ul> |
| | <ul> <li>Persons who have been prescribed PAP therapy by a physician</li> </ul> |
| | <ul> <li>Persons who are existing nasal mask or sub-nasal mask users with</li> <li>≥3 months of use prior to enrolment in the clinical trial</li> </ul> |
| | <ul> <li>Persons who are compliant with PAP therapy for ≥4 hours per night<br/>for ≥70% of nights for a 14-day period within 30 days prior to<br/>enrolment in the clinical trial</li> </ul> |
| | Persons who are fluent in spoken and written English |
| | Persons who possess the capacity to provide informed consent |
| | Exclusion criteria: |
| | Persons who are intolerant to PAP therapy |
| | <ul> <li>Persons who possess, or suffer from, anatomical or physiological<br/>conditions which make PAP therapy inappropriate</li> </ul> |
| | <ul> <li>Persons who are required to use PAP therapy for &gt;12 hours per day<br/>or for extensive periods, not including sleep or naps</li> </ul> |
| | <ul> <li>Persons who are trying to get pregnant, are pregnant, or think they may be pregnant</li> </ul> |
| | <ul> <li>Persons who have an IPAP pressure of &gt;30 cmH<sub>2</sub>O if on BPAP</li> </ul> |
| | <ul> <li>Persons who use a PAP therapy device for the delivery of<br/>medicines, except supplemental oxygen</li> </ul> |
| | <ul> <li>Persons who use a PAP therapy device that does not possess data<br/>recording capabilities to capture AHI and a numerical indicator of<br/>leak that is accessible to the investigation site</li> </ul> |

F&P , 2023

| Information | Details |
|---|---|
| Number of Subjects | Recruitment target for patient participants: Between 40 and45 |
| Duration of Clinical<br>Investigation | |
| Total number of visits in clinical investigation | |
| Background and Rationale | The F&P |
| Phase of Development | As per ISO-14155:2020, 'Annex I', the F&P mask is considered in the pivotal stage of device development. |
| Study Design | clinical investigation. |
| Study Hypotheses | Patient Participant Primary hypothesis: The F&P |



F&P , US, 2023

| Information | Petaile |
|---|---|
| Information | Details |
| Clinical Investigation<br>Objective(s) | Patient Participant: |
| Objective(s) | To evaluate the performance, comfort, stability and reliability of the F&P mask among patient participants using PAP therapy, with regards to patient participant views on overall experience, satisfaction and acceptance. |
| Sponsor Details | <u> </u> |
| Sponsor Name | |
| Sponsor Representative Name | |
| Sponsor Address | |
| Co-ordinating Investigator Name(s) | |
| Co-ordinating Investigator<br>Professional Position(s) | |
| Co-ordinating Investigator<br>Business / Clinic / Hospital<br>Name | Fisher & Paykel Healthcare |
| Co-ordinating Investigator<br>Business / Clinic / Hospital<br>Address | 15 Maurice Paykel Place East Tamaki Auckland 2013 New Zealand |
| Investigator Details | |
| Principal Investigator Name | |
| Principal Investigator<br>Professional Position | |
| Principal Investigator Clinic | |
| Principal Investigator Clinic<br>Address | |

&P , US, 2023

Doc. No:

Revision: A

| Information | Details |
|--------------------------------------------------------------------|---------|
| Co-ordinating Investigator Name(s) | |
| Co-ordinating Investigator<br>Professional Position(s) | |
| Co-ordinating Investigator<br>Business / Clinic / Hospital<br>Name | |
| Investigation Site details | |
| Investigation site | |
| Investigation site address | |

# 2. Identification and Description of the Investigational Device

| Information | Details |
|---|---|
| Summary Description of Medical Device | mask used for the delivery of positive airway pressure to the upper airways. |
| Details concerning the manufacturer of the investigational device | |
| Name/Number of model | F&P |
| Description of how traceability shall be achieved | Product accountability logs will be used to keep a record for product traceability. |
| Intended purpose of the investigational device | The F&P mask is intended to be used as a patient interface in a non-invasive positive airway pressure (PAP) therapy system to deliver pressurized air from the breathing tube to the patient's upper airway. |
| Populations and indications for which the investigational device is intended | The patients are intended to be adults weighing ≥30 kg or 66 pounds. |

&P , US, 2023

Doc. No:
Revision:

| Information | Details |
|---|---|
| Description of the investigational device | |
| Summary of the necessary training and experience needed to use investigational device | Training sessions covering the investigational product and protocol for the investigation sites and PI's will be conducted prior to the investigation starting. The investigational device will be fitted to the subjects by a trained F&P staff member. |
| Description of any specific medical or surgical procedures involved in the use of the clinical device. | N/A |
| Reference to IB and IFU | The IB can be found for this clinical investigation |

# 3. Justification for the Design of the clinical investigation

### 3.1. Synopsis

The investigation is a prospective, non-randomized, non-blinded study. This clinical investigation is designed to validate and confirm the overall performance and acceptability of the F&P

provides positive airway pressure (PAP) therapy for existing patients which is equivalent to the treatment provided by their usual mask.

are commonly used as part of PAP therapy, both in clinical settings and in-home environments for the treatment of various respiratory conditions, including obstructive sleep apnea (OSA).

### 3.2. Literature Review

A full description of PAP therapy and the associated conditions which can be effectively treated PAP is located

P , US, 2023

Doc. No:

Revision:

A

Positive airway pressure (PAP) and non-invasive ventilation (NIV) are common treatments used in chronic care to assist in airway management for several respiratory conditions present in both adults and adolescents, including obstructive sleep apnea (OSA), obesity hypoventilation syndrome (OHS), among others. The prevalence of these conditions, as well as others, continues to rise as the prevalence of noncommunicable diseases, such as obesity, increase across many parts of the world<sup>8,9</sup> Historically, invasive methods of ventilation were required to maintain airway patency, but this is often associated with significant long-term medical complications as well as increased susceptibility to other conditions<sup>10</sup>. Non-invasive methods, if appropriate for a patient, are now more appealing to practicing physicians, especially if treatment is administered in a non-clinical setting, such as the home.



PAP therapy was first described in 1981<sup>11</sup> for the treatment of OSA, a form or sleep-disordered breathing (SDB) characterized by upper airway collapse during sleep. PAP therapy is now a well-established, effective, and the clinically preferred treatment for OSA, helping resolve many of the primary markers of disease severity<sup>3</sup>. It has evolved to include a variety of modes including auto-titrating positive airway pressure (APAP), bilevel positive airway pressure (BPAP), and continuous positive airway pressure (CPAP), as well as comfort features such as humidification and expiratory relief (ER) which improve uptake and long-term adherence among those prescribed with the treatment<sup>3</sup>. PAP therapy is delivered through a system of components which includes a flow generator, breathing tube, and interface, sometimes with the addition of a humidifier or mask accessory.

It is generally accepted that PAP therapy:

- Is safe to use among adults with OSA
- Reduces Apnea-Hypopnea Index (AHI) and excessive daytime sleepiness (EDS) among adults with OSA
- Reduces AHI among adults with OHS
- . In the form of APAP and CPAP are equally efficacious for treating adults with OSA

PAP and NIV therapies are still considered the most effective and reliable treatment options for those with OSA and OHS, despite advancements in alternative treatments such as oral appliances (OA) and surgical interventions to remodel structures at the back of the throat such as tonsillectomies or uvulopalatopharyngoplasties 10,12. Professional organizations continue to recommend PAP or NIV therapy, where applicable and appropriate, over alternative treatments. In order to deliver effective therapy, the components which make up the treatment system must work harmoniously. While the effective pressure is determined by a practicing physician, the machine which generates flow must accurately and consistently deliver required prescribed constant or fluctuating pressures.

F&P US, 2023

Doc. No:

Revision:

A

The interface should provide an effective seal over the face to minimize leak, a factor which significantly impacts the sleep quality and level of comfort experienced by patients, as well as their long-term tolerance and adherence to treatment<sup>3,13</sup>. While there are a significant number of benefits to using PAP and NIV therapies for the relevant indications, both also come with some risks to the patient. These include potential sleep disruption, facial irritation, mandibular pain, internal trauma, anxiety sensitivity, abdominal discomfort, physiological compromise, facial discomfort, facial dryness, mucosal congestion, and facial inflammation. However, manufactures of medical devices which deliver PAP and NIV therapies can address a number of these side effects with improving design and functionality. This may involve the incorporation of humidification and ER technologies in machines, or the use of comfortable and non-irritating materials for interfaces

| 3.3. Pre-Clinical Testing |
|---|
| PAP therapy is a treatment designed to be administered to humans. |
| a series of bench tests is conducted on the investigational product to ensure it is safe and will perform as expected when used on human subjects. |
| product to ensure it is sale and will perform as expected when used on human subjects. |
| 3.4. Previous Clinical trial |
| The main objective of the F&P mask is to develop a |
| . The F&P |
| The F&P |




F&P , US, 2023

| F&P Servision 3.5. Justification for Administration There is an ongoing need for advancement in design and technology for PAP therapy is specifically as a means of improving comfort for patients and encouraging log-term administration. Benefits and Risks of the investigational device, clinical indical investigation 4.1. Anticipated benefits 4.2. Risks associated with participation in the clinical investigation. AP therapy is currently one of the least invasive and most widely recommended treatments erves as the generally accepted state of the art within the field of sleep and respiratory medical investigatory medical investigation and respiratory medical investigation. | nasks on the mar |
|---|---|
| 3.5. Justification for Administration There is an ongoing need for advancement in design and technology for PAP therapy in specifically as a means of improving comfort for patients and encouraging log-term administration. Benefits and Risks of the investigational device, clinical indical investigation 4.1. Anticipated benefits 4.2. Risks associated with participation in the clinical investigation. AP therapy is currently one of the least invasive and most widely recommended treatments. | nasks on the mar<br>erence to treatm |
| There is an ongoing need for advancement in design and technology for PAP therapy in specifically as a means of improving comfort for patients and encouraging log-term advancement in design and technology for PAP therapy in specifically as a means of improving comfort for patients and encouraging log-term advancements and Risks of the investigational device, clinical indexident clinical investigation 4.1. Anticipated benefits 4.2. Risks associated with participation in the clinical investigation are the reapy is currently one of the least invasive and most widely recommended treatments. | erence to treatm |
| Benefits and Risks of the investigational device, clinical nd clinical investigation 4.1. Anticipated benefits 4.2. Risks associated with participation in the clinical investigation AP therapy is currently one of the least invasive and most widely recommended treatments | erence to treatm |
| 4.1. Anticipated benefits 4.2. Risks associated with participation in the clinical investigation AP therapy is currently one of the least invasive and most widely recommended treatments | procedure |
| 4.2. Risks associated with participation in the clinical investigation AP therapy is currently one of the least invasive and most widely recommended treatments | |
| 4.2. Risks associated with participation in the clinical investigation AP therapy is currently one of the least invasive and most widely recommended treatments | |
| AP therapy is currently one of the least invasive and most widely recommended treatments | |
| rves as the generally accepted state of the art within the field of sleep and respiratory med | |
| ceptability of risk associated with PAP therapy devices, interfaces, accessories, and supp | |
| chnology for delivering treatment to the target population are shared, and is appropriate, a | the benefits of |
| AP therapy outweigh most risks. | |
| 4.3. Possible interactions with concomitant medical treatments | |
| 4.4. Steps that will be taken to control or mitigate risks | |
| The F&P | |
| | _ |

PAP therapy is considered standard treatment for those diagnosed with OSA,

RP US, 2023

Doc. No: Revision: A

# 5. Objectives & Hypotheses of the clinical investigation

# 5.1. **Objectives** 5.1.1. Patient participant objective To evaluate the performance, comfort, usability, stability, and reliability of the F&P mask among participants using PAP therapy, with regards to participant views on overall experience, satisfaction, and acceptance. 5.2. **Hypotheses** 5.2.1. Patient participant hypothesis Primary hypothesis: The F&P mask is effective in providing adequate PAP therapy, or treatment comparable to that provided by the usual mask used by participants, for managing a respiratory condition during in-home use. Secondary hypothesis: The F&P mass mask presents an acceptable safety profile when used by participants with PAP therapy for the management of a respiratory condition during in-home use.

F&P N, US, 2023 


Revision: A

&P US, 2023

Doc. No: Revision:

A

## **5.4.** Methods and Timing for assessing, recording and analysing variables

| Fisher&Paykel HEALTHCARE | | | |
|---|---|---|---|
| F&P | US, 2023 | Doc. No:<br>Revision: | A |
| | assessing clinical investigation vari | ables and arrange | ments for |
| monitoring maintenance and o | calibration | | |
| 5.7. Investigation sites | | | |
| This is a single-site clinical investigatio | on. | ŀ | |
| 5.7.1. Definition of completion of c | _ | | |
| - Phase 1 will be complete who | en the patient participants have comple | eted | |
| - The participants will be offere | ed to participate in Phase 2, | | |
| | e(s) and comparator(s) | | |
| o.o. mivesugational devic | scia, and comparatoria, | | |

, US, 2023

Doc. No: Revision: Δ



## 6. Participants

### 6.1.1. Inclusion criteria for participants selection

F&P following inclusion and exclusion criteria.

### Inclusion criteria for patient participant:

- Persons who are ≥22 years of age
- Persons who weigh ≥66 pounds (or 30 kg)
- Persons who have been prescribed PAP therapy by a physician
- Persons who are existing nasal mask or sub-nasal mask users with ≥3 months of use prior to enrolment in the clinical trial
- Persons who are compliant with PAP therapy for ≥4 hours per night for ≥70% of nights for a 14-day period within 30 days prior to enrolment in the clinical trial
- Persons who are fluent in spoken and written English
- Persons who possess the capacity to provide informed consent

| _ |
|---|

### **6.1.2.** Exclusion criteria for participants selection

### **Exclusion criteria for patient participant:**

- Persons who are intolerant to PAP therapy
- Persons who possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate

&P US, 2023

Doc. No: Revision:



- Persons who are required to use PAP therapy for >12 hours per day or for extensive periods, not including sleep or naps
- Persons who are trying to get pregnant, are pregnant, or think they may be pregnant
- Persons who have an IPAP pressure of >30 cmH<sub>2</sub>O if on BPAP
- Persons who use a PAP therapy device for the delivery of medicines, except supplemental oxygen
- Persons who use a PAP therapy device that does not possess data recording capabilities to capture
   AHI and a numerical indicator of leak that is accessible to the investigation site

| 6.1.3. Criteria and procedures for patients withdrawal / lost to follow-up | |
|---|---|
| Participants will be informed that they have the right to withdraw from the clinical investigation at any time, | |
| without prejudice or compromise to their medical care, and are not obliged to state their reasons. | |
| | 8 |
| | I |
| | ı |
| | l |

The PI may withdraw a participant at any time for the following reasons:

- Protocol violation
- · Safety concerns
- Serious illness
- AEs

| 6.1.4. | Point of Enrolment |
|--------|--------------------|

| Fish | ner&Paykel<br>ALTHCARE | | | | | |
|---|---|---|---|---|---|---|
| | F&P | | , US, 2023 | | Doc. No: Revision: | |
| | 9 | | | | | |
| | _ | | | | | |
| • | | | | | <u> </u> | |
| | Detient menticinents on | manlatina Dhaca 4 wi | II b | Alex aliminal image | - <b>4</b> ; <b>4</b> ; | |
| | Patient participants co | mpleting Phase 1 Wil | ii be participating in | the clinical inves | stigation | |
| | Clayton Sleep Institute | will recruit up to 45 p | atient participants fo | or the F&P Nova | Nasal clinical | investigation |
| | , | | | | | g |
| | | | | | | - |
| There | is no intention to recru | it individuals in vulne | rable populations. | | | |
| 7. | Procedures | | _ | | | |
| The p | rotocol of this clinical ir | vestigation is summa | arized | | | |
| | | | | | | <u>-</u> |


&P US, 2023

Doc. No: Revision:

Α




RP US, 2023



F&P , US, 2023

Doc. No: Revision: A

## 7.1.1. Clinical-Investigation Procedures



| Do. No. Revision: A C. Procedures that will be carried out Below are the activities | Fishe | er& <b>Paykel</b><br>LTHCARE | | | Pag | e 28 of 69 |
|---|---|---|---|---|---|---|
| D. Procedures that will be carried out | | | F&P | US, 2023 | | |
| D. Procedures that will be carried out | | | | | Revision. A | |
| D. Procedures that will be carried out | | | | | | |
| D. Procedures that will be carried out | | | | <u> </u> | | |
| D. Procedures that will be carried out | | | | | | |
| Procedures that will be carried out | C. | | | | | |
| Procedures that will be carried out | | | | | | |
| Procedures that will be carried out | | | | | | |
| Procedures that will be carried out | | | | | | |
| Procedures that will be carried out | D | | | | | |
| E. | ٥. | | | | | |
| E. E. | | | | | | |
| E. E. | | | | | | |
| E. E. | | Procedures th | nat will be carried out | | | |
| E. | | | | | | |
| E. | | | | | | |
| E. | | | | | | |
| E. | | | | | | |
| E. | | | | | | |
| E. E. | | | | | | |
| | E | | | | | |
| Below are the activities | | | | | | |
| Below are the activities | | | | | | |
| Delow are the activities | | Polovy or a H- | activities | | | |
| | | Delow are the | a activities | | | |

| Fisher HEA | er&Paykel | | | | | |
|---|---|---|---|---|---|---|
| | | F&P | | US, 2023 | Doc. No:<br>Revision: | A |
| | | | | | Revision. | A |
| F. | | | | | | |
| | Below are th | | | | | |
| G. | | | | | | |
| О. | | | | | | |
| | Below are th | e activities | | | | |
| Н. | | | | | | |
| | Procedures t | that will be carri | ed out | | | |
| | | | | | | _ |



## 7.2. Roles and Responsibilities



US, 2023 Doc. No: Revision: A

| Fisher & Paykel HEALTHCARE | | | |
|---|---|---|---|
| | F&P | US, 2023 | Doc. No: Revision: A |
| Participants will be | ational prod<br>factory. | on of their enrolment in the clini | cal investigation cal investigation may be terminated if |
| The following is red | quired | | |
| ' | | | |
| ' | | | |
| | onitoring Plan | | |
| Fisher & Pa | ykel Healthcare (F&P) | will appoint | |

| | F&P | US, 2023 | Doc. No: Revision: A |
|--------------|---------|----------|----------------------|
| Responsib | ilities | | |
| Specific tas | | | |
| | | _ | |

| Fisher & Paykel HEALTHCARE | | | | |
|---|---|---|---|---|
| HEALTHCARE | | | Doc Not | 1 agc 34 01 03 |
| | F&P | , US, 2023 | Doc. Not Revision: | A |
| | | | T COVIDION. | |

| Fisher & Paykel<br>HEALTHCARE | F&P | , US, 2023 | Doc. No:<br>Revision: | |
|---|---|---|---|---|
| | | | | • |
| Statistic | al Design and A | Analysis | | |

&P US, 2023

Doc. No: Revision:

A

| | 8.1.1. Safety Data |
|---|---|
| Adverse even | ts (AE) and serious adverse events (SAE) will be captured as part of the clinical investigation |
| 8.2. | Sample size calculation and justification |
| Patient Partic | |
| Between 40 a | nd 45 patient participants will be recruited for this clinical investigation. |



F&P Doc. No:
Revision: A

| _ |
|---|




F&P , US, 2023

Doc. No: Revision: A

| | All partic | ipants who consent and who use the investigational product |
|---|---|---|
| 9. | Data | Management |

| | | | | Page 39 of |
|---|---|---|---|---|
| | F&P | , US, 2023 | Doc. No:<br>Revision: | A |
| | | | TROVIDION. | |
| T. C | | " ( | | |
| The following | persons have auth | ority to amend the CIP: | | |
| Deviatio | ons from clini | ical investigation pl | lan (CIP) | |
| Deviation | ons from clini | ical investigation pl | lan (CIP) | |
| | | ical investigation pl | | |

Revision:

## 12. Device Accountability



| Fish | ner&Paykel<br>althcare | | | |
|---|---|---|---|---|
| | F&P | US, 2023 | Doc. No:<br>Revision: | A |
| | The F&P the requirements | clinical investigation is being co | nducted in the USA and ther | efore must mee |
| 14. | Informed Cons | ent Process | | |

E&P US, 2023

Doc. No: Revision: Δ

## 15. Adverse Events, Adverse device effects and device deficiencies



16.

US, 2023

Doc. No: Revision:

| • |
|---|
| Δ |

| Suspension or premature termination of clinical investigation |
|---|
| Participants will be followed up with throughout the duration of their enrolment in the clinical investigation |





## 18. Regulatory and Other References





F&P US, 2023 

Doc. No: Revision: A




F&P US, 2023

Doc. No:

Revision:

A

| _ |
|---|
| _ |
| _ |
| _ |
| _ |
| _ |

F&P US, 2023 


Revision: A

| Fisher&Paykel | | | | |
|---------------|-----|------------|-----------------------|---------------|
| | F&P | , US, 2023 | Doc. No:<br>Revision: | A |
| | _ | _ | | |




F&P , US, 2023

Doc. No:

Revision: A

| i |
|---|

| F&P Doc. No: Revision: A | <b>Fisher</b> & <b>Paykel</b><br>HEALTHCARE | | | |
|---|---|---|---|---|
| Revision. A | | F&P | IIS 2023 | |
| | | 1 0.1 | , 00, 2020 | Revision: A |

| Fisher&Paykel<br>HEALTHCARE | | | | |
|---|---|---|---|---|
| | F&P | , US, 2023 | Doc. No:<br>Revision: | A |

| Fisher & Paykel |
|-----------------|
| HEALTHCARE |


&P , US, 2023

Doc. No: Revision:

Α

































This document is not controlled when printed.

Refer to Fisher & Paykel Healthcare intranet for current revision.